CLINICAL TRIAL: NCT01873261
Title: Neurally Adjusted Ventilatory Assist (NAVA) Versus Pressure Support in Pediatric Acute Respiratory Failure - Pilot Study
Brief Title: NIV NAVA Versus NIV-PS in Pediatric Patients - Pilot Study
Acronym: NINAVAPed
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Ignacio Galicia, Dr, Hospital Universitario La Paz
Other Study IDs: HULP-PI-3750
Record Dates: First submitted 2013-02-19; First posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Acute Respiratory Failure
Keywords: Neurally Adjusted Ventilatory Assist; Pediatric Acute Respiratory Failure; non-invasive ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This pilot study will be an observational no randomize study in which the NiNAVAped protocol will be applied solely to the NIV NAVA arm.

DETAILED DESCRIPTION:
This pilot study will be an observational no randomize study in which the NiNAVAped protocol will be applied solely to the NIV NAVA arm.

Every PICU will have to include 3 patients in the Pilot study before starting the clinical trial, which means that the pilot study will involve a maximum of 60 patients.

Should the Pilot study reveal deficiencies in the NiNAVAped design, the protocol would be improved accordingly.

There will be a specific consent document during the Pilot study. The Pilot study will be published in a scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 1 month age to 18 years
* Moderate/severe Pediatric Acute Respiratory failure of any origin evaluated after a period of respiratory stabilization (aspiration of secretions, physiotherapy, oxygen and nebulized therapy) when the attending pediatric intensive care physician believes that the patient is likely to require endotracheal intubation (ETI).
* Non intubated
* Admitted to the PICU
* Minimally agitated/sedated: between -2 and +2 on the Richmond agitation-sedation scale (Table 2)

Exclusion Criteria:

1. Patients younger than 1 month or older than 18 year
2. Patients who need immediate endotracheal intubation: i.e.: Severe ARF with signs of exhaustion
3. Facial trauma/burns
4. Recent facial, upper way, or upper gastrointestinal tract surgery excepting gastrostomy for feeding
5. Fixed obstruction of the upper airway
6. Inability to protect airway
7. Life threatening hypoxemia defined as SpaO2 <90% with FiO2 > 0.8 on hi-flow oxygen.
8. Hemodynamic instability: refractory at volume expansion >60 ml/kg and dopamine >10 mcg/kg/min
9. Impaired consciousness defined as Glasgow coma scale < 10.
10. Bowel obstruction.
11. Untreated pneumothorax.
12. Poor short term prognosis (high risk of death in the next 3 months)
13. Known esophageal problem (hiatal hernia, esophageal varicosities)
14. Active upper gastro-intestinal bleeding or any other contraindication to the insertion of a NG tube.
15. Neuromuscular disease
16. Vomiting
17. Cough or gag reflex impairment.
18. Cyanotic congenital heart disease.
19. Complete absence of cooperation
20. This patient has been included (randomized) previously in the study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children from 1 month to 18 years admitted to the PICU with moderate/severe acute respiratory failure minimally sedated/agitated
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Avoiding endotracheal intubation using non-invasive ventilation | During non invasive ventilation, an average of 2-3 days.
  The primary endpoint of this study is avoiding endotracheal intubation (ETI) (and conventional mechanical ventilation (MV)) using non-invasive ventilation (NIV). It is defined as no need for ETI (and MV) for at least 48h after the withdrawal of NIV.

SECONDARY OUTCOMES:
Length (days) of endotracheal intubation (conventional mechanical ventilation) after NIV | During mechanical ventilation after NIV
Length (days) of PICU stay after NIV | After NIV
  The patients will be follow up after NIV during the PICU stay, and average of two weeks
Length (days) hospital stay after NIV | After NIV
  The patients will be follow up after NIV during hospital stay, an average of 2-3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kacmarek, PhD RRT FCCM, Study Director — Massachusetts General Hospital, Boston, USA; Jesús Villar, MD, PhD, Principal Investigator — Hospital Universitario Dr. Negrin
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Cheifetz IM. Invasive and noninvasive pediatric mechanical ventilation. Respir Care. 2003 Apr;48(4):442-53; discussion 453-8. PMID 12667269
- [Background] Kendirli T, Kavaz A, Yalaki Z, Ozturk Hismi B, Derelli E, Ince E. Mechanical ventilation in children. Turk J Pediatr. 2006 Oct-Dec;48(4):323-7. PMID 17290566
- [Background] Al-Mutairi SS, Al-Deen JS. Non-invasive positive pressure ventilation in acute respiratory failure. An alternative modality to invasive ventilation at a general hospital. Saudi Med J. 2004 Feb;25(2):190-4. PMID 14968216
- [Background] L'HerE, Moriconi M, Texier F, Bouquin V, Kaba L, Renault A, Garo B, Boles JM. Non-invasive continuous positive airway pressure in acute hypoxaemic respiratory failure--experience of an emergency department. Eur J Emerg Med. 1998 Sep;5(3):313-8. PMID 9827833
- [Background] Bernet V, Hug MI, Frey B. Predictive factors for the success of noninvasive mask ventilation in infants and children with acute respiratory failure. Pediatr Crit Care Med. 2005 Nov;6(6):660-4. doi: 10.1097/01.pcc.0000170612.16938.f6. PMID 16276332
- [Background] Calderini E, Chidini G, Pelosi P. What are the current indications for noninvasive ventilation in children? Curr Opin Anaesthesiol. 2010 Jun;23(3):368-74. doi: 10.1097/ACO.0b013e328339507b. PMID 20440111
- [Background] Keenan SP, Sinuff T, Cook DJ, Hill NS. Does noninvasive positive pressure ventilation improve outcome in acute hypoxemic respiratory failure? A systematic review. Crit Care Med. 2004 Dec;32(12):2516-23. doi: 10.1097/01.ccm.0000148011.51681.e2. PMID 15599160
- [Background] Essouri S, Durand P, Chevret L, Haas V, Perot C, Clement A, Devictor D, Fauroux B. Physiological effects of noninvasive positive ventilation during acute moderate hypercapnic respiratory insufficiency in children. Intensive Care Med. 2008 Dec;34(12):2248-55. doi: 10.1007/s00134-008-1202-9. Epub 2008 Aug 19. PMID 18712350
- [Background] Breatnach C, Conlon NP, Stack M, Healy M, O'Hare BP. A prospective crossover comparison of neurally adjusted ventilatory assist and pressure-support ventilation in a pediatric and neonatal intensive care unit population. Pediatr Crit Care Med. 2010 Jan;11(1):7-11. doi: 10.1097/PCC.0b013e3181b0630f. PMID 19593246
- [Background] Biban P, Serra A, Polese G, Soffiati M, Santuz P. Neurally adjusted ventilatory assist: a new approach to mechanically ventilated infants. J Matern Fetal Neonatal Med. 2010 Oct;23 Suppl 3:38-40. doi: 10.3109/14767058.2010.510018. PMID 20828233
- [Background] Munoz-Bonet JI, Flor-Macian EM, Brines J, Rosello-Millet PM, Cruz Llopis M, Lopez-Prats JL, Castillo S. Predictive factors for the outcome of noninvasive ventilation in pediatric acute respiratory failure. Pediatr Crit Care Med. 2010 Nov;11(6):675-80. doi: 10.1097/PCC.0b013e3181d8e303. PMID 20308933